CLINICAL TRIAL: NCT06777303
Title: Efficacy of Locally Applied Nano-Curcumin and Nano-Hyaluronic Acid as an Adjunct to Scaling and Root Planing in the Treatment of Periodontitis Patients
Brief Title: Efficacy of Nano-Curcumin and Nano-Hyaluronic Acid as an Adjunct to Scaling and Root Planing in the Treatment of Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A05010240M
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (-ve control group) SRP alone (Active Comparator): are treated with scaling and root planning alone
  Interventions: Procedure: scaling and root planning
- group 2 ( +ve control group) SRP + chitosan nano-particles LDD (Active Comparator): patients are treated with SRP in addition to chitosan nano-particles as an adjunct local drug delivery.
  Interventions: Drug: chitosan nano-particles
- group 3 ( experimental group 1) SRP + curcumin loaded on chitosan nano-particles (Experimental): patients are treated with SRP in addition to curcumin loaded on chitosan nano-particles as an adjunct local drug delivery.
  Interventions: Drug: curcurmin loaded on chitosan nano-particles
- group 4 ( experimental group 2) SRP + hyaluronic acid loaded on chitosan nano-particles (Experimental): patients are treated with SRP in addition to hyaluronic-acid loaded on chitosan nano-particles as an adjunct local drug delivery.
  Interventions: Drug: hyaluronic acid loaded on chitosan nano-particles

INTERVENTIONS:
Drug: curcurmin loaded on chitosan nano-particles — the formulation of curcumin and incorprating it with chitosan nano-particles will increase the absorption rate in the gingival sulcus
  Arms: group 3 ( experimental group 1) SRP + curcumin loaded on chitosan nano-particles
Drug: hyaluronic acid loaded on chitosan nano-particles — the formulation of hyaluronic acid and incorprating it with chitosan nano-particles will increase the absorption rate in the gingival sulcus
  Arms: group 4 ( experimental group 2) SRP + hyaluronic acid loaded on chitosan nano-particles
Procedure: scaling and root planning — the -ve control group in the study
  Arms: group 1 (-ve control group) SRP alone
Drug: chitosan nano-particles — the +ve control group in the study
  Arms: group 2 ( +ve control group) SRP + chitosan nano-particles LDD

SUMMARY:
to evaluate Efficacy of Locally Applied Nano-Curcumin and Nano-Hyaluronic Acid as an Adjunct to Scaling and Root Planing in the Treatment of Periodontitis patients

Materials and methods: forty patients (n=40) were selected from the Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mansoura University, The participants forty patients are classified into four groups:

* Group1 : (-ve control group): SRP alone
* Group2: (+ve control group): SRP+ chitosan Nano-particles
* Group3: SRP + Curcumin-coated chitosan Nano-particles
* Group4: SRP+ hyaluronic acid -coated chitosan Nano-particle

All Patients will undergo Phase I therapy, which includes scaling and root planing using ultrasonic tips and gracey curettes. Additionally, mechanical oral hygiene instructions will be provided, and participants will be advised to refrain from using any mouthwash throughout the duration of the study.

Furthermore, patients within groups 2 to 4 will be subjected to an extra measure involving the application of the respective gel associated with their designated group. The gel will be administered on a weekly basis for duration of five weeks.

Clinical indices (plaque index (PI), gingival index (GI), clinical attachment level (CAL), and probing depth (PD)). Laboratory assessment will be done at baseline and final assessment( after 3 months) . tess will be for antioxdiant levels and TNF alpha

* Total anti-oxidant capacity(T-AOC) using Assay kit50T
* TNF alpha using ELISA Kit (96T)

DETAILED DESCRIPTION:
Inclusion criteria:

Patients who are systemically healthy Patient exhibiting periodontal pocket depths (PD) ≤5mm presence of clinical attachment loss (CAL) between 1-4mm cooperative individuals capable of adhering to mechanical oral hygiene instructions Patients who agreed on both written and verbal consent to participate in the study.

6

o Exclusion criteria: patients with recent history of periodontal treatment (within the last 3 months) patients with recent use of antibiotic (within the past 3 months, pregnant or lactating women, individuals who are malnourished and taking vitamin supplements, Patients who regularly use mouthwashes.

Method of gel application: a blunt 2ml syringe will be used to administer the gel sub-gingivally until the pocket is filled

Cervicular fluid collection :

This is done at baseline and after 12 weeks

* Insert absorbent paper points gently into the gingival crevice at the sulcus or pocket depth.
* Allow the absorbent material to remain in the crevice for a specific duration (1 minute) to enable the collection of gingival crevicular fluid.
* Carefully retrieve the paper points from the gingival crevice, ensuring that the collected fluid is preserved on the material.
* Place the paper points in eppendorf tubes
* Handle the samples with care to prevent contamination and promptly transport them to the laboratory for further analysis. If necessary, samples may undergo centrifugation to separate cells and debris from the fluid.

Periodontal assessment:

The following periodontal indices will be assessed at baseline, and after 12 weeks o Plaque Index according to Silness P. Loe H 1964

* Gingival Bleeding Index/Bleeding On Probing(BOP) according to Ainamo & Bay 1975
* Probing pocket depth (PPD) is measured from free gingival margin to base of the pocket.
* Clinical attachment loss (CAL) is measured from cemento-enemal junction to base of the pocket.

the determination of the sample size was guided by reference of similar articles. . Employing G power for the calculation, the sample size was determined with a 0.676 effect size, a two-tailed test, α error set at 0.05, and a power of 0.8, resulting in a total calculated sample size of 10 individuals in each group.

Pretreatment period Participants were informed about the purpose of the study and screened for eligibility. They also were informed about the treatment received and the steps done, including non-surgical treatment and gel application with the associated risks, possible effects, and other treatment options available. The participants understood this explanation in broad terms according to the rules of the ethical committee of the Faculty of Dentistry, Mansoura University. Additionally, they acknowledged that they would be required to attend the periodic recall visits and that they are legally competent to give written informed consent before performing any required steps.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are systemically healthy
* Patient exhibiting periodontal pocket depths (PD) ≤5mm
* presence of clinical attachment loss (CAL) between 1-4mm
* cooperative individuals capable of adhering to mechanical oral hygiene instructions
* Patients who agreed on both written and verbal consent to participate in the study.

Exclusion Criteria:

* patients with recent history of periodontal treatment (within the last 3 months)
* patients with recent use of antibiotic (within the past 3 months)
* pregnant or lactating women,
* individuals who are malnourished and taking vitamin supplements,
* Patients who regularly use mouthwashes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth reduction | 12 weeks
  pocket depth is calculated using a UNC 15 perio probe to calculate the distance between the base of the pocket to the free gingival margin

SECONDARY OUTCOMES:
plaque index | 12 weeks
  according to Silness P. Loe H 1964
clinical attachment gain | 12 weeks
  measured from cemento-enemal junction to base of the pocket
Gingival Bleeding Index | 12 weeks
  according to Ainamo & Bay 1975
o Total anti-oxidant capacity(T-AOC) | 12 weeks
  laboratory investigation using Assay kit50T
tumor necrosis factor alpha (TNF alpha) | 12 weeks
  laboratory investigation using ELISA Kit (96T)

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided